CLINICAL TRIAL: NCT06366438
Title: A Randomized Controlled Trial of Two Universal Programs for Parents of Teenagers: ABC (Face-to-face) vs. Parentweb (Online)
Brief Title: A Trial of Two Universal Programs for Parents of Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Forster, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ABC vs Parentweb
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Mental Disorder; Adolescent Behavior; Adolescent Development; Parent-Child Relations; Parenting
Keywords: Parenting; Randomized controlled trial; Parent-Child relations; Prevention; Universal
MeSH Terms: conditions — Mental Disorders; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of the three arms upon allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABC-teen (Experimental): The ABC-teen is a universal parenting program where two trained leaders meet parents meet in groups (10-15 parents) at four occasions (2.5 hours each). One or two follow-up meetings are also offered. The themes that are covered during the meetings include: spending time together, communication, parental stress management and emotion regulation, and problem solving/conflict resolution.
  Interventions: Behavioral: ABC-teen
- ParentWeb (Experimental): ParentWeb is an online-based program where parents individually work with material online (text, images, clips, quizzes), while they receive support from a parent guide through asynchronous text messages. The program includes four main modules that are expected to be covered in eight weeks. The themes of the modules include: spending time together, communication, problem solving/conflict resolution, and keeping in touch while letting go of control.
  Interventions: Behavioral: ParentWeb
- Wait-List (No Intervention): The parents will be on a six months wait-list control group.

INTERVENTIONS:
Behavioral: ABC-teen — See above
  Arms: ABC-teen
Behavioral: ParentWeb — See above
  Arms: ParentWeb

SUMMARY:
Parent training programs in groups and over internet can help parents improve their interaction and communication with their children. There is however a lack knowledge of how programs work for parents of teenagers, as most studies have concerned younger children. Furthermore, most studies have been conducted on programs for selective populations with elevated risk. The aim of this study was to investigate the effectiveness of two universal preventive parenting programs for teenagers: The group-based program 'ABC-teen' and the online-based 'ParentWeb'. Both programs aim to strengthen the parent-adolescent relationship and reduce negative communication. The programs are developed in Sweden with content based on other established parenting programs (e.g., Comet, Incredible Years, the Triple P). The aim of the present study was to evaluate the effects of the the two programs, with adolescent mental health as primary outcome. Several secondary outcome measures concerning parenting and parent-adolescent relationship were also collected. Parents were randomized to ABC-teen, ParentWeb or a 6 months Wait-List control. Parent- and adolescent ratings were collected at baseline, after 4 and after 12 months. All data collection has now been completed and the next step is to process and analyze the data.

DETAILED DESCRIPTION:
BACKGROUND:

Despite the development of psychological treatments in recent decades, mental health disorders remain a main cause of disease, functional impairments, and deaths of adolescents across the world. UNICEF estimated that globally, over 13 percent of adolescents 10-19 live with a mental disorder. Moreover, suicide is the fifth most common cause of death for adolescents in the same age-span and the fourth most prevalent cause for adolescents 15-19 years old. Reports also show that youth mental illness have increased in recent years. Psychological treatments seems not enough to combat this negative development; preventive efforts are needed.

Family experiences can be a target of prevention given the strong impact on young peoples' current and future mental health. The quality of the parent-child relationship impacts health quality throughout life. Also, adverse experiences related to family and parenting dysfunction is one of the main predictors of mental ill-health. While adolescence is a period of increased independence, parents remain one of the most important people in the young person's life. A link between parenting factors during adolescence and anxiety and depression, which constitutes 40% of diagnosed adolescent mental disorders, is established. Parenting factors linked to depression and anxiety include low warmth, inter-parental conflict, over-involvement, and aversiveness.

Decades of research support the health benefits of parent training programs that help parents interact and communicate with their children, including face-to-face programs delivered in groups and internet-based programs. However, most studies have concerned children below 13 years of age. Given the impact of parenting factors during adolescence on mental health, it is important to investigate how parenting programs work for parents of adolescents.

Parenting programs on different prevention levels are needed to maximize the benefit on public health. However, most studies have concerned indicated/selected prevention or treatments. Outcomes have mostly concerned symptom reduction. To prevent health problems at a population scale, more studies are needed of how parenting programs benefit the general population (i.e., universal prevention). The general population includes those who do not presently experience clinical problems, but where future issues may be prevented through strengthening health-promoting factors (e.g., family relationships).

PURPOSE AND RESEARCH QUESTIONS:

The aim of this study is to assess the effectiveness of two universal preventive parenting programs for teenagers: ABC-teen and ParentWeb. A version of the ABC program for children 3-12 years old has been evaluated in a randomized controlled trial, but so far no study has investigated ABC-teen. Likewise, a longer version of the ParentWeb targeting a selected group of parents with elevated levels of conflict with their adolescents has been published, but no study on the universal version of ParentWeb. The effects of the programs will be evaluated both in comparison to each other and to a Wait-List control. Both programs aim to strengthen the parent-adolescent relationship and reduce negative communication.

1. What are the programs' effect on adolescent and parental mental health?
2. What are the programs' effect on parenting behaviors and parental self-efficacy?
3. What are the programs' effect on the relationship between parents and adolescents?
4. What are the programs' effect on school adjustment?
5. What are the programs' effect on the adolescents' use of tobacco, alcohol and drugs?
6. To what extent do the parents experience participation in the programs' as feasible and satisfying?

   Research question 1-6 will be reported in the main paper from the project, while the following research questions will be reported in following papers.
7. Are there predictors and moderators of program effects (e.g., demographic variables and variables related to implementation/adherence)?
8. What are the health economic outcomes of the programs?

METHOD:

Participants:

The sample consisted of 1247 families (1327 parents and 471 adolescents) from the general population, from 58 sites in 52 municipalities across Sweden. The participants were recruited through local advertisements in schools or online municipality channels. Parents who were interested were referred to a website with additional information and a consent form. All members in a family (parents and adolescents) were invited to contribute to the data collection in the study (questionnaires).

Design:

The study is a multi-site randomized controlled trial. Parents were randomized to ABC-teen, ParentWeb or a 6 months Wait-List control. After recruitment, participants responded to baseline measurements and were subsequently randomized to one of the three study conditions. The randomization was conducted centrally by the researchers, but with separate randomization list for each site (generated at randomize.org). The researchers then informed a local coordinator at the site about participants' allocation. Parents and adolescents who were included at baseline were invited to answer follow-up questionnaires after 4 and 12 months. The wait-list control group parents were invited to participate in either ABC-teen or ParentWeb (their choice) after 6 months. Thus, at the 12 month follow-up, analyses of program effects will be restricted to comparisons between the programs.

Sample size calculation:

As the effects of universal interventions are generally small, a relatively large study group was required for adequate statistical power, also considering that drop-out can be substantial in multi-site studies. For a statistical power of 80%, 200 participating families will be needed to detect small differences in effect size (Cohen's d = .20) with alpha = 0.05. Since the randomization was unbalanced (2-1-1 in ABC-teen, ParentWeb, and wait list), an additional 200 families had to be recruited to reach at least 200 in each condition (i.e., 400 in ABC-teen, 200 in ParentWeb, and 200 in the wait list). This means that a total of 800 families with complete data were needed for the study. To account for dropout, an additional 447 families were recruited. Actual n:s in each condition at each measurement point were as follows at the completion of data collection: ABC-teen - 669 (baseline), 520 (4 month), 458 (12 month); ParentWeb - 297 (baseline), 209 (4 month), 168 (12 month); Wait list - 281 (baseline), 210 (4 month).

Statistical analyses:

Linear Mixed Modeling (LMM) will be used for analyzing the effects of the programs (questions 1-5) in two steps: First, effects at 4 month will be analyzed comparing each of the program to the wait list control. Second, the two programs will be compared to each other at 4 and 12 month. For questions 6, t-tests will be conducted to investigate mean differences between the two program conditions. For question 7, LMM-analyses will be conducted with predictors and moderators entered into the equations, to test if they have (differential) effects on the slope of adolescent mental health and parenting variables from baseline to 12 month follow-up. For question 8, two different health economic analyses will be conducted - one analyzing the cost of health gains in terms of quality of life (by mapping scores from the SDQ to preference-based utility values), and another analyzing the cost of health gains in terms of reduced mental illness (recovered cases). All analyses will be conducted according to Intention-to-treat (primary results), as well as per protocol (sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* A caregiver or another adult who live part- or full-time with at least one adolescent 13-19 years old.

Exclusion Criteria:

* The family had an ongoing contact (treatment or assessment) concerning a child or adolescent within the psychiatry, social services, primary psychiatric care, habilitation, or equivalent services.
* Health or language deficiencies that make it difficult to respond to questionnaires or participate in group or online parent support.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1247 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
The Strength and Difficulties Questionnaire (SDQ) | Pre (0 month), 4 months, 12 months
  Measures adolescent mental health. Rated by parents and adolescents. The scale consists of five sub-scales and a supplement. In this study, the Total problem scale will be used as primary outcome measure. The Total problem scale consists of the sum of the following four sub-scales: Hyperactivity, Emotional problems, Conduct problems, and Peer problems. The range of the Total problem scale is 0 to 60 points, where higher scores indicate more problems.
Patient Health Questionnaire (PHQ-9) | Pre (0 month), 4 months, 12 months
  Measures parental mental health (specifically depression). Rated by parents. The range of the scale is 0 to 27 points, where higher scores indicates more depressive symptoms.
Parental stress scale (PSS) | Pre (0 month), 4 months, 12 months
  Measures parental mental health (specifically parental stress). Rated by parents. The range of the scale is 0 to 32 points, where higher scores indicate more stress.
General Anxiety Disorder Scale (GAD-7) | Pre (0 month), 4 months, 12 months
  Measures parental mental health (specifically anxiety). Rated by parents. The range of the scale is 0 to 21, where higher scores indicate more symptoms of anxiety.

SECONDARY OUTCOMES:
Conflict scale | Pre (0 month), 4 months, 12 months
  Measures the relationship between the parent and the adolescent. The scale measure the frequency of everyday conflicts between the parent and the adolescent. A number of typical conflicts are listed and the participants are asked to rate how frequently they have occurred on a likert scale from 0 (never) to 3 (often). Rated by parents and adolescents.
Adult Child Relationship Scale (ACRS) | Pre (0 month), 4 months, 12 months
  Measures the relationship between the parent and the adolescent (specifically expressions of warmth and closeness in the relationship). It includes 6 items (e.g., "If my teenager is upset, he/she turns to me for support") which are rated on a likert scale from 0 (I do not agree at all) to 4 (I agree completely). Rated by parents and adolescents.
Adolescents' openness scale | Pre (0 month), 4 months, 12 months
  Measures the relationship between the parent and the adolescent (specifically teenagers openness with their parents). It includes 6 items (e.g., "Does your teenager tell you which peers he/she has hanged out with if he/she has been out?"), which are rated on a likert scale from 0 (never) to 4 (almost always). Rated by parents and adolescents.
Brief Family Relationship Scale | Pre (0 month), 4 months, 12 months
  Measures the relationship in the family as a whole. It includes 15 items (e.g., "In our family we really get along well with each other."), which are rated on a likert scale from 1 (Do not agree at all) to 20 (Agrees completely). Rated by parents.
Positive and Negative Parenting Behaviors | Pre (0 month), 4 months, 12 months
  Measures parent behaviors. The scale consists of 4 items that has been used in a large scale dissemination study of ABC for children 3-12 years (e.g., "How often have you been spending time or doing something nice together with your teenager the past two weeks?" and "How often have you been nagging on your teenager the past two weeks?"). The items are rated on a likert scale from 1 (Never) to 7 (Several times a day). Rated by parents.
Me as a Parent | Pre (0 month), 4 months, 12 months
  Measures parental self-efficacy. The scale consists of 16 items (e.g., "I am satisfied with the way I am able to emotionally support my teenager"), which are rated on a likert scale from 0 (Do not agree at all) to 4 (Agree to a high extent). Rated by parents.
Conflict Resolution Efficacy | Pre (0 month), 4 months, 12 months
  Measures parental self-efficacy (specifically self-efficacy regarding management of conflicts). The scale is connected to the Conflict Scale described above. For each type of conflict that at least has occurred to some extent during the past two weeks (e.g. "Conflicts regarding screen-time"), the following sub-question appears: "How did you manage to handle those conflicts?". The sub-questions are rated on a likert scale from 1 (Badly) to 10 (Good). Rated by parents.
School Adjustment Scale | Pre (0 month), 4 months, 12 months
  Measures the school adjustment. The scale consists of four items from an annual survey used nationally by school districts in Sweden (e.g., "I find the school work interesting"). Each item is rated on a likert scale from 0 (I do not agree at all) to 3 (I agree completely). Rated by parents and adolescents.
Stockholmsenkaten | Pre (0 month), 4 months, 12 months
  The scale consists of 9 items from a yearly school survey used in the school district of Stockholm to measures adolescent use of tobacco, alcohol and drugs. The data from the measure can both used as dichotomous outcomes (Ever used tobacco/alcohol/drugs? YES/NO), but also as a continuous outcome since the frequency of use (if any) also is measured. When used as a continuous outcome, the scale includes the three sub scales: Tobacco (range 0-6 points), Alcohol (range 0-25 points), and Drugs (range 0-12 points). For all sub scales, higher values indicate higher frequency of use.
Satisfaction Questionnaire | At 4- and 12 month follow-ups.
  Measures parents satisfaction with participation in the parenting programs. The scale consists of four items concerning the extent to which the parents experience that the program has led to improvements, has helped them in general, and how likely it is that they would recommend it to a friend. Each item is rated on a likert scale from 0 (Not at all) to 3 (Very much). Rated by parents.
Attendance and engagement measures | At 4- and 12 month follow-ups.
  Measures attendance and engagement, which indirectly indicates feasibility. Questions regarding attendance/completion of each meeting/module and regarding homework completion, for both the responding parent as well as co-parents. Rated by parents (and staff).

OTHER OUTCOMES:
Demographics | Pre (0 month)
  Questions to assess family background and living conditions. Not outcome measures, but to be used in analyses of predictors and moderators.
Organizational and therapist factors | Pre (0 month)
  Questions about organizational and personnel factors (e.g. group leader background). Not outcome measures, but to be used in analyses of predictors and moderators. Rated by group leaders.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, PhD, Principal Investigator — Karolinska Institutet
Locations (58):
- Sweden (58):
  - Bromma stadsdel, Bromma
  - Danderyd kommun, Danderyd
  - Ovanåkers kommun, Edsbyn
  - Farsta stadsdel, Farsta
  - Göteborgs kommun, Gothenburg
  - Götene kommun, Götene
  - Värmdö kommun, Gustavsberg
  - Hallsbergs kommun, Hallsberg
  - Haninge kommun, Handen
  - Hägersten-Älvsjö stadsdel, Hägersten
  - Tellusborgsskolan, Hägersten
  - Aspuddens skola, Hägersten
  - Hässelby Vällingby stadsdel, Hässelby
  - Höörs kommun, Höör
  - Huddinge kommun, Huddinge
  - Järfälla kommun, Jakobsberg
  - Skarpnäck stadsdel, Johanneshov
  - Enskede Årsta Vantör stadsdel, Johanneshov
  - Karlsborgs kommun, Karlsborg
  - Kungälvs kommun, Kungälv
  - Upplands-Bro kommun, Kungsängen
  - Leksands kommun, Leksand
  - Lidingö kommun, Lidingö
  - Lidköpings kommun, Lidköping
  - Lilla Edets kommun, Lilla Edet
  - Lindesbergs kommun, Lindesberg
  - Linköpings kommun, Linköping
  - Lomma kommun, Lomma
  - Lunds kommun, Lund
  - Mariestads kommun, Mariestad
  - Sigtuna kommun, Märsta
  - Nacka kommun, Nacka
  - Norrköpings kommun, Norrköping
  - Norrtälje kommun, Norrtälje
  - Nynäshamns kommun, Nynäshamn
  - Sävsjö kommun, Sävsjö
  - Skärholmen stadsdel, Skärholmen
  - Skellefteå kommun, Skellefteå
  - Skövde kommun, Skövde
  - Sollentuna kommun, Sollentuna
  - Stenungsunds kommun, Stenungsund
  - Kungsholmen stadsdel, Stockholm
  - Norra Real, Stockholm
  - Norrmalm stadsdel, Stockholm
  - Östermalm stadsdel, Stockholm
  - Södermalm stadsdel, Stockholm
  - MFJ Hammarby Sjöstad, Stockholm
  - Sundbybergs stad, Sundbyberg
  - Sundsvalls kommun, Sundsvall
  - Täby kommun, Täby
  - Tidaholms kommun, Tidaholm
  - Töreboda kommun, Töreboda
  - Trelleborgs kommun, Trelleborg
  - Botkyrka kommun, Tumba
  - Vallentuna kommun, Vallentuna
  - Växjö kommun, Vaxjo
  - Vällingbyskolan, Vällingby
  - Gotlands kommun, Visby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Florean IS, Dobrean A, Pasarelu CR, Georgescu RD, Milea I. The Efficacy of Internet-Based Parenting Programs for Children and Adolescents with Behavior Problems: A Meta-Analysis of Randomized Clinical Trials. Clin Child Fam Psychol Rev. 2020 Dec;23(4):510-528. doi: 10.1007/s10567-020-00326-0. Epub 2020 Sep 8. PMID 32897527
- [Background] Bausback KB, Bunge EL. Meta-analysis of parent training programs utilizing behavior intervention technologies. Soc Sci. 2021;10(10):367. https://doi.org/10.3390/socsci1010 0367 21.
- [Background] Kaminski JW, Claussen AH. Evidence Base Update for Psychosocial Treatments for Disruptive Behaviors in Children. J Clin Child Adolesc Psychol. 2017 Jul-Aug;46(4):477-499. doi: 10.1080/15374416.2017.1310044. Epub 2017 May 1. PMID 28459280
- [Background] Leijten P, Gardner F, Melendez-Torres GJ, van Aar J, Hutchings J, Schulz S, Knerr W, Overbeek G. Meta-Analyses: Key Parenting Program Components for Disruptive Child Behavior. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):180-190. doi: 10.1016/j.jaac.2018.07.900. Epub 2018 Nov 26. PMID 30738545
- [Background] Ulfsdotter M, Enebrink P, Lindberg L. Effectiveness of a universal health-promoting parenting program: a randomized waitlist-controlled trial of All Children in Focus. BMC Public Health. 2014 Oct 18;14:1083. doi: 10.1186/1471-2458-14-1083. PMID 25326710
- [Background] Wetterborg D, Enebrink P, Lonn Rhodin K, Forster M, Risto E, Dahlstrom J, Forsberg K, Ghaderi A. A pilot randomized controlled trial of Internet-delivered parent training for parents of teenagers. J Fam Psychol. 2019 Oct;33(7):764-774. doi: 10.1037/fam0000541. Epub 2019 Jun 17. PMID 31204818
- [Background] Stewart-Brown SL, Fletcher L, Wadsworth ME. Parent-child relationships and health problems in adulthood in three UK national birth cohort studies. Eur J Public Health. 2005 Dec;15(6):640-6. doi: 10.1093/eurpub/cki049. Epub 2005 Aug 10. PMID 16093299
- [Background] Green JG, McLaughlin KA, Berglund PA, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and adult psychiatric disorders in the national comorbidity survey replication I: associations with first onset of DSM-IV disorders. Arch Gen Psychiatry. 2010 Feb;67(2):113-23. doi: 10.1001/archgenpsychiatry.2009.186. PMID 20124111
- [Background] Yap MB, Pilkington PD, Ryan SM, Jorm AF. Parental factors associated with depression and anxiety in young people: a systematic review and meta-analysis. J Affect Disord. 2014 Mar;156:8-23. doi: 10.1016/j.jad.2013.11.007. Epub 2013 Nov 18. PMID 24308895
- [Background] Racine N, McArthur BA, Cooke JE, Eirich R, Zhu J, Madigan S. Global Prevalence of Depressive and Anxiety Symptoms in Children and Adolescents During COVID-19: A Meta-analysis. JAMA Pediatr. 2021 Nov 1;175(11):1142-1150. doi: 10.1001/jamapediatrics.2021.2482. PMID 34369987
- [Background] United Nations Children's Fund [UNICEF], The State of the World's Children 2021: On My Mind - Promoting, protecting and caring for children's mental health, UNICEF, New York, October 2021.
- [Background] Holmes EA, Ghaderi A, Harmer CJ, Ramchandani PG, Cuijpers P, Morrison AP, Roiser JP, Bockting CLH, O'Connor RC, Shafran R, Moulds ML, Craske MG. The Lancet Psychiatry Commission on psychological treatments research in tomorrow's science. Lancet Psychiatry. 2018 Mar;5(3):237-286. doi: 10.1016/S2215-0366(17)30513-8. No abstract available. PMID 29482764
- [Background] Sanders MR, Divan G, Singhal M, Turner KMT, Velleman R, Michelson D, Patel V. Scaling Up Parenting Interventions is Critical for Attaining the Sustainable Development Goals. Child Psychiatry Hum Dev. 2022 Oct;53(5):941-952. doi: 10.1007/s10578-021-01171-0. Epub 2021 May 4. PMID 33948778